CLINICAL TRIAL: NCT00394004
Title: Exploring Decision Making of Hispanics and African Americans With HIV/AIDS Participating in Clinical Trials
Brief Title: Decision-Making of Hispanics and African-Americans With HIV/AIDS Participating in Clinical Trials
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070015; 07-CC-0015
Record Dates: First submitted 2006-10-28; First posted 2006-10-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-26

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: Decision Making; Health Disparities; Hispanic; African-American; Clinical Trials; HIV Positive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; HIV Seropositivity

SUMMARY:
This study will use focus groups and in-depth individual interviews to explore factors that influence the decision of Hispanics and African-Americans with HIV/AIDS to participate in a research study.

HIV-positive Hispanic and African-American patients 18 years of age and older who are enrolled in an NIH HIV/AIDS protocol may be eligible for Part 1, Part 2, or both parts of this study, as follows:

Part 1 - Focus group

Focus group participants of from six to ten people are interviewed together during a one-time, 2-hour tape-recorded session to explore how they arrived at their decision to enroll in a research study. The group discussion is led by a moderator and a facilitator. Before the session begins, participants complete questionnaires that include information about their age, race, ethnicity, education and social support. Hispanic participants also complete a questionnaire about language preference. At the end of the focus group, participants are offered to be interviewed individually, as described below.

Part 2 - In-depth interview

An investigator conducts a one-on-one in-depth interview with the participant while a second person observes and tape records the interview. The interview may take from 1 1/2 to 2 hours to complete. Participants who were not in a focus group are asked to complete questionnaires as described in Part 1 above.

DETAILED DESCRIPTION:
The realities of health disparities are well documented. The HIV/AIDS epidemic is a health crisis for African Americans and a serious threat to the Hispanic Community. In 2003, African Americans accounted for 50% of the new HIV/AIDS cases. According to the U.S. Census Bureau, Census 2000 Brief, African Americans/Blacks make up 12.9% of the U.S. population and account for 40% of the 929,985 estimated AIDS cases. The U. S. Census Bureau also reports as of May 2001 Hispanics account for 12.5% of the population. In 2002, the Centers for Disease Control (CDC) reported that Hispanics accounted for 13% of the new cases with an increase of 26% since 1999. As the numbers indicate, HIV/AIDS is a serious concern to both African Americans and Hispanics.

Additionally there is an underrepresentation of Hispanics and African Americans in clinical trials. It is critical that Hispanics and African Americans with HIV/AIDS be included in clinical trials. Minority underrepresentation in clinical trials prohibits generalizability of results and is of significant concern.

In this study, we propose examining the decision making processes of Hispanics and African Americans with HIV/AIDS around their decision to enter a clinical trial in an effort to develop a future instrument to measure decision making in this population. This is a descriptive, exploratory mixed methods study designed to examine the decision-making process among a convenience sample of minority patients who are enrolled in active HIV/AIDS protocols.

Through focus groups and in-depth interviews, participants will be asked about the factor(s) that influence their decision to participate in research. By asking the participants directly, we may gain a better understanding of their decision-making process. Obtaining these data may provide strategies for facilitating inclusion of Hispanics and African Americans with HIV/AIDS into clinical trials.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients enrolled in at least one active NIH HIV/AIDS protocol.
  2. Age greater than or equal to 18 years.
  3. Willingness and capacity to provide informed consent.
  4. Self-identifying as Hispanic/Latino or African American/Black.
  5. Be HIV-positive.
  6. Willing to have comments recorded on audiotape.

EXCLUSION CRITERIA:

1. Age less than 18 years.
2. Self-identifying as other than Hispanic/Latino or African American/Black.
3. Patients only enrolled in the Natural History HIV Protocol, 95-I-0072, Clinical Virologic and Immunologic Evaluation and Monitoring of Patients with Known or Suspected HIV Infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-10-26; Study Completion 2011-04-26

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Acevedo MC. The role of acculturation in explaining ethnic differences in the prenatal health-risk behaviors, mental health, and parenting beliefs of Mexican American and European American at-risk women. Child Abuse Negl. 2000 Jan;24(1):111-27. doi: 10.1016/s0145-2134(99)00121-0. PMID 10660014
- [Background] Alderete E, Vega WA, Kolody B, Aguilar-Gaxiola S. Lifetime prevalence of and risk factors for psychiatric disorders among Mexican migrant farmworkers in California. Am J Public Health. 2000 Apr;90(4):608-14. doi: 10.2105/ajph.90.4.608. PMID 10754977
- [Background] Allen M, Israel H, Rybczyk K, Pugliese MA, Loughran K, Wagner L, Erb S. Trial-related discrimination in HIV vaccine clinical trials. AIDS Res Hum Retroviruses. 2001 May 20;17(8):667-74. doi: 10.1089/088922201750236942. PMID 11429107